CLINICAL TRIAL: NCT01332188
Title: A Single Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Efficacy of Three Different Concentrations of Cetirizine (0.05%, 0.1%, and 0.24%) Ophthalmic Solution Versus Vehicle in the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge Model (CAC)
Brief Title: Efficacy of AC-170 for the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge (CAC) Model
Acronym: AC-170
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-100-0004
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC-170 0.05% (Experimental)
  Interventions: Drug: AC-170 0.05%
- AC-170 0.1% (Experimental)
  Interventions: Drug: AC-170 0.1%
- AC-170 0.24% (Experimental)
  Interventions: Drug: AC-170 0.24%
- AC-170 0% (Placebo Comparator)
  Interventions: Drug: AC-170 0%

INTERVENTIONS:
Drug: AC-170 0.05% — 1 drop in each eye at 3 separate times during a 21 day period
  Arms: AC-170 0.05%
Drug: AC-170 0.1% — 1 drop in each eye at 3 separate times during a 21 day period
  Arms: AC-170 0.1%
Drug: AC-170 0.24% — 1 drop in each eye at 3 separate times during a 21 day period
  Arms: AC-170 0.24%
Drug: AC-170 0% — 1 drop in each eye at 3 separate times during a 21 day period
  Arms: AC-170 0%

SUMMARY:
The purpose of this study is to evaluate the efficacy of different concentrations of AC-170 compared to vehicle in the prevention of the signs and symptoms of allergic conjunctivitis in the conjunctival allergen challenge (CAC) Model.

ELIGIBILITY:
Inclusion Criteria:

* Positive bilateral conjunctival allergen challenge (CAC) reaction

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to the study enrollment or during the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one site in the US.
Pre-assignment Details: 101 subjects were enrolled, 7 subjects discontinued, and 94 subjects completed the study. The 101 subjects that met all inclusion criteria and none of the exclusion criteria were randomized to receive AC-170 0.05%, AC-170 0.1%, AC-170 0.24% or AC-170 0%.
  Note: All solutions were "early formulations" and not the final to-be-marketed formulation.
Period: Overall Study
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Started | 25 | 26 | 25 | 25
Completed | 23 | 25 | 21 | 25
Not Completed | 2 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0% | Total
Number analyzed (Participants) | 25 | 26 | 25 | 25 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.58) | 43.1 (13.5) | 38.9 (12.53) | 38.1 (14.12) | 41.4 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 10 | 14 | 56
  Male | 8 | 11 | 15 | 11 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 5 | 16
  Not Hispanic or Latino | 22 | 21 | 22 | 20 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 24 | 25 | 24 | 23 | 96
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 25 | 25 | 101

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  3 minutes post-CAC | 1.91 (0.924) | 2.00 (0.771) | 1.65 (0.963) | 2.48 (0.540)
  5 minutes post-CAC | 2.01 (1.019) | 2.04 (0.889) | 1.74 (0.843) | 2.55 (0.550)
  7 minutes post-CAC | 1.86 (0.907) | 1.87 (0.913) | 1.75 (0.910) | 2.27 (0.777)

2. Primary Outcome: Ocular Itching at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  3 minutes post-CAC | 1.99 (0.849) | 1.78 (0.873) | 1.90 (0.804) | 2.24 (0.575)
  5 minutes post-CAC | 2.00 (0.711) | 1.92 (0.883) | 2.17 (0.819) | 2.24 (0.686)
  7 minutes post-CAC | 1.77 (0.774) | 1.78 (0.988) | 1.97 (0.833) | 2.08 (0.702)

3. Primary Outcome: Ocular Itching at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  3 minutes post-CAC | 1.05 (0.804) | 0.84 (0.800) | 0.91 (0.810) | 1.94 (0.870)
  5 minutes post-CAC | 1.19 (0.778) | 1.09 (0.941) | 1.07 (0.840) | 2.09 (0.850)
  7 minutes post-CAC | 1.01 (0.789) | 1.07 (0.929) | 0.97 (0.843) | 1.94 (0.893)

4. Primary Outcome: Conjunctival Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.62 (0.634) | 1.59 (0.624) | 1.45 (0.489) | 1.79 (0.359)
  15 minutes post-CAC | 1.68 (0.606) | 1.65 (0.711) | 1.61 (0.545) | 1.91 (0.426)
  20 minutes post-CAC | 1.63 (0.696) | 1.58 (0.721) | 1.56 (0.634) | 1.88 (0.403)

5. Primary Outcome: Conjunctival Redness at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.43 (0.635) | 1.38 (0.668) | 1.71 (0.628) | 1.70 (0.505)
  15 minutes post-CAC | 1.63 (0.617) | 1.59 (0.663) | 1.85 (0.608) | 1.90 (0.489)
  20 minutes post-CAC | 1.61 (0.617) | 1.54 (0.677) | 1.79 (0.713) | 1.76 (0.575)

6. Primary Outcome: Conjunctival Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.44 (0.663) | 1.45 (0.812) | 1.66 (0.718) | 1.88 (0.541)
  15 minutes post-CAC | 1.81 (0.670) | 1.67 (0.821) | 1.83 (0.680) | 1.96 (0.589)
  20 minutes post-CAC | 1.83 (0.648) | 1.67 (0.868) | 1.79 (0.717) | 1.97 (0.622)

7. Secondary Outcome: Ciliary Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.47 (0.708) | 1.53 (0.758) | 1.34 (0.684) | 1.81 (0.527)
  15 minutes post-CAC | 1.60 (0.707) | 1.65 (0.842) | 1.52 (0.732) | 1.99 (0.523)
  20 minutes post-CAC | 1.60 (0.703) | 1.65 (0.878) | 1.53 (0.788) | 1.95 (0.573)

8. Secondary Outcome: Ciliary Redness at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  7 minutes post-CAC: number analyzed (Participants) | 23 | 25 | 25 | 25
  7 minutes post-CAC | 1.36 (0.730) | 1.22 (0.686) | 1.50 (0.633) | 1.55 (0.582)
  15 minutes post-CAC: number analyzed (Participants) | 23 | 25 | 25 | 25
  15 minutes post-CAC | 1.49 (0.596) | 1.47 (0.723) | 1.74 (0.716) | 1.77 (0.544)
  20 minutes post-CAC: number analyzed (Participants) | 23 | 25 | 25 | 25
  20 minutes post-CAC | 1.50 (0.617) | 1.47 (0.701) | 1.65 (0.736) | 1.65 (0.599)

9. Secondary Outcome: Ciliary Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 24
units on a scale
  7 minutes post-CAC | 1.24 (0.689) | 1.24 (0.867) | 1.27 (0.858) | 1.67 (0.628)
  15 minutes post-CAC | 1.59 (0.749) | 1.51 (0.861) | 1.64 (0.669) | 1.77 (0.661)
  20 minutes post-CAC | 1.65 (0.647) | 1.52 (0.952) | 1.73 (0.622) | 1.79 (0.644)

10. Secondary Outcome: Episcleral Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.68 (0.602) | 1.74 (0.690) | 1.57 (0.497) | 1.90 (0.439)
  15 minutes post-CAC | 1.81 (0.639) | 1.77 (0.757) | 1.69 (0.605) | 2.02 (0.484)
  20 minutes post-CAC | 1.80 (0.629) | 1.73 (0.797) | 1.69 (0.647) | 1.97 (0.458)

11. Secondary Outcome: Episcleral Redness at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.53 (0.590) | 1.37 (0.681) | 1.73 (0.616) | 1.80 (0.505)
  15 minutes post-CAC | 1.72 (0.585) | 1.63 (0.700) | 1.90 (0.657) | 2.00 (0.505)
  20 minutes post-CAC | 1.70 (0.579) | 1.60 (0.688) | 1.87 (0.696) | 1.85 (0.530)

12. Secondary Outcome: Episcleral Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 1.52 (0.644) | 1.49 (0.782) | 1.64 (0.744) | 1.93 (0.508)
  15 minutes post-CAC | 1.86 (0.652) | 1.73 (0.803) | 1.98 (0.698) | 2.01 (0.575)
  20 minutes post-CAC | 1.91 (0.577) | 1.72 (0.861) | 1.88 (0.644) | 2.04 (0.598)

13. Secondary Outcome: Chemosis at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Chemosis was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of chemosis score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.71 (0.553) | 0.58 (0.406) | 0.53 (0.292) | 0.72 (0.532)
  15 minutes post-CAC | 0.93 (0.557) | 0.70 (0.545) | 0.60 (0.354) | 0.99 (0.575)
  20 minutes post-CAC | 0.92 (0.644) | 0.72 (0.583) | 0.71 (0.460) | 1.00 (0.650)

14. Secondary Outcome: Chemosis at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Chemosis was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of chemosis score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.68 (0.478) | 0.52 (0.279) | 0.55 (0.298) | 0.68 (0.399)
  15 minutes post-CAC | 0.87 (0.612) | 0.64 (0.396) | 0.77 (0.433) | 0.81 (0.532)
  20 minutes post-CAC | 0.90 (0.647) | 0.71 (0.419) | 0.84 (0.572) | 0.90 (0.568)

15. Secondary Outcome: Chemosis at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Chemosis was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of chemosis score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  7 minutes post-CAC: number analyzed (Participants) | 23 | 25 | 25 | 24
  7 minutes post-CAC | 0.49 (0.232) | 0.43 (0.293) | 0.54 (0.277) | 0.74 (0.427)
  15 minutes post-CAC | 0.74 (0.423) | 0.52 (0.314) | 0.79 (0.456) | 0.80 (0.554)
  20 minutes post-CAC | 0.71 (0.403) | 0.53 (0.363) | 0.76 (0.399) | 0.88 (0.555)

16. Secondary Outcome: Eyelid Swelling at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Eyelid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of eyelid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.6 (0.75) | 0.8 (0.66) | 0.8 (0.66) | 0.9 (0.71)
  15 minutes post-CAC | 0.7 (0.79) | 0.9 (0.75) | 0.8 (0.54) | 1.1 (0.86)
  20 minutes post-CAC | 0.6 (0.76) | 0.8 (0.73) | 0.7 (0.56) | 1.0 (0.85)

17. Secondary Outcome: Eyelid Swelling at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Eyelid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of eyelid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.7 (0.60) | 0.7 (0.54) | 0.9 (0.68) | 0.7 (0.74)
  15 minutes post-CAC | 0.8 (0.70) | 0.8 (0.73) | 0.9 (0.82) | 0.9 (0.82)
  20 minutes post-CAC | 0.8 (0.69) | 0.8 (0.76) | 0.9 (0.72) | 0.9 (0.85)

18. Secondary Outcome: Eyelid Swelling at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Eyelid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of eyelid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.4 (0.56) | 0.5 (0.70) | 0.5 (0.49) | 0.7 (0.81)
  15 minutes post-CAC | 0.5 (0.68) | 0.6 (0.65) | 0.6 (0.65) | 0.8 (0.89)
  20 minutes post-CAC | 0.5 (0.71) | 0.6 (0.58) | 0.5 (0.49) | 0.7 (0.84)

19. Secondary Outcome: Tearing at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Tearing was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of tearing score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.0 (1.07) | 0.8 (0.72) | 0.6 (0.51) | 0.6 (0.67)
  15 minutes post-CAC | 0.8 (0.89) | 0.5 (0.64) | 0.7 (0.65) | 0.9 (0.82)
  20 minutes post-CAC | 0.7 (0.85) | 0.4 (0.63) | 0.7 (0.62) | 0.9 (0.97)

20. Secondary Outcome: Tearing at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Tearing was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of tearing score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.0 (0.78) | 0.7 (0.61) | 0.6 (0.75) | 0.8 (0.71)
  15 minutes post-CAC | 1.1 (0.79) | 0.6 (0.54) | 0.7 (0.66) | 0.8 (0.82)
  20 minutes post-CAC | 1.0 (0.77) | 0.5 (0.53) | 0.7 (0.72) | 0.7 (0.84)

21. Secondary Outcome: Tearing at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Tearing was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of tearing score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.7 (0.74) | 0.5 (0.49) | 0.3 (0.56) | 0.6 (0.64)
  15 minutes post-CAC | 0.5 (0.66) | 0.5 (0.50) | 0.4 (0.50) | 0.6 (0.64)
  20 minutes post-CAC | 0.5 (0.60) | 0.4 (0.47) | 0.2 (0.33) | 0.6 (0.90)

22. Secondary Outcome: Rhinorrhea at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Rhinorrhea was assessed by the patient on a 0-4 scale (0=none to 4=severe). Rhinorrhea score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.1 (1.26) | 0.4 (0.49) | 0.7 (0.99) | 0.7 (0.80)
  15 minutes post-CAC | 1.2 (1.01) | 0.6 (0.77) | 1.1 (1.04) | 1.0 (1.12)
  20 minutes post-CAC | 1.3 (1.14) | 0.7 (0.80) | 1.1 (1.05) | 1.1 (1.24)

23. Secondary Outcome: Rhinorrhea at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Rhinorrhea was assessed by the patient on a 0-4 scale (0=none to 4=severe). Rhinorrhea score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.1 (1.28) | 0.6 (0.65) | 0.8 (0.90) | 0.7 (0.69)
  15 minutes post-CAC | 1.1 (1.29) | 0.7 (0.69) | 1.2 (0.91) | 1.0 (0.84)
  20 minutes post-CAC | 1.2 (1.28) | 0.6 (0.70) | 1.0 (0.71) | 0.8 (0.90)

24. Secondary Outcome: Rhinorrhea at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Rhinorrhea was assessed by the patient on a 0-4 scale (0=none to 4=severe). Rhinorrhea score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.6 (1.20) | 0.2 (0.41) | 0.3 (0.58) | 0.6 (0.82)
  15 minutes post-CAC | 0.9 (1.25) | 0.4 (0.65) | 0.5 (0.75) | 0.8 (0.87)
  20 minutes post-CAC | 0.8 (1.23) | 0.4 (0.71) | 0.5 (0.68) | 0.6 (0.70)

25. Secondary Outcome: Nasal Pruritus at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Nasal Pruritus was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.6 (0.91) | 0.2 (0.37) | 0.5 (0.65) | 0.4 (0.71)
  15 minutes post-CAC | 0.6 (0.91) | 0.4 (0.65) | 0.7 (0.80) | 0.8 (1.01)
  20 minutes post-CAC | 0.7 (0.99) | 0.6 (0.91) | 0.6 (0.65) | 0.8 (1.13)

26. Secondary Outcome: Nasal Pruritus at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Nasal Pruritus was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.7 (0.93) | 0.4 (0.64) | 0.4 (0.58) | 0.4 (0.82)
  15 minutes post-CAC | 0.7 (1.03) | 0.4 (0.58) | 0.8 (0.93) | 0.6 (0.99)
  20 minutes post-CAC | 0.5 (0.90) | 0.5 (0.65) | 0.6 (0.82) | 0.7 (0.85)

27. Secondary Outcome: Nasal Pruritus at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Nasal Pruritus was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.4 (0.99) | 0.2 (0.37) | 0.3 (0.56) | 0.4 (0.65)
  15 minutes post-CAC | 0.4 (0.84) | 0.3 (0.56) | 0.2 (0.44) | 0.4 (0.58)
  20 minutes post-CAC | 0.4 (0.95) | 0.4 (0.64) | 0.3 (0.66) | 0.4 (0.65)

28. Secondary Outcome: Ear or Palate Pruritus at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.4 (0.87) | 0.4 (0.57) | 0.3 (0.74) | 0.5 (0.87)
  15 minutes post-CAC | 0.9 (1.09) | 0.8 (0.90) | 0.5 (0.77) | 1.0 (1.10)
  20 minutes post-CAC | 0.8 (1.11) | 0.9 (0.91) | 0.8 (0.93) | 1.2 (1.31)

29. Secondary Outcome: Ear or Palate Pruritus at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.6 (0.89) | 0.3 (0.46) | 0.4 (0.76) | 0.5 (0.96)
  15 minutes post-CAC | 0.7 (0.96) | 0.6 (0.65) | 0.7 (0.98) | 0.8 (1.19)
  20 minutes post-CAC | 0.8 (1.11) | 0.7 (0.74) | 0.7 (0.90) | 0.7 (1.07)

30. Secondary Outcome: Ear or Palate Pruritus at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.6 (0.99) | 0.2 (0.52) | 0.3 (0.56) | 0.4 (0.76)
  15 minutes post-CAC | 08 (0.95) | 0.4 (0.76) | 0.3 (0.58) | 0.7 (1.07)
  20 minutes post-CAC | 0.7 (1.01) | 0.5 (0.77) | 0.3 (0.58) | 0.7 (1.07)

31. Secondary Outcome: Nasal Congestion at Onset of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Nasal Congestion was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Congestion score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 1.2 (0.99) | 0.5 (0.65) | 0.8 (1.18) | 0.8 (0.78)
  15 minutes post-CAC | 1.4 (1.04) | 0.6 (0.76) | 1.0 (1.19) | 1.2 (0.85)
  20 minutes post-CAC | 1.5 (1.05) | 0.8 (0.99) | 1.0 (1.14) | 1.3 (1.21)

32. Secondary Outcome: Nasal Congestion at Duration of Action (24 Hours Post-dose)
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Nasal Congestion was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Congestion score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 25 | 25
units on a scale
  7 minutes post-CAC | 0.9 (0.97) | 0.6 (0.58) | 0.8 (0.80) | 0.7 (0.69)
  15 minutes post-CAC | 1.2 (0.98) | 0.6 (0.58) | 1.2 (0.94) | 1.1 (0.83)
  20 minutes post-CAC | 1.2 (1.00) | 0.6 (0.65) | 1.1 (1.04) | 1.2 (0.88)

33. Secondary Outcome: Nasal Congestion at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Nasal Congestion was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Congestion score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
units on a scale
  7 minutes post-CAC | 0.7 (1.05) | 0.4 (0.58) | 0.4 (0.59) | 0.8 (0.78)
  15 minutes post-CAC | 1.1 (1.08) | 0.5 (0.65) | 0.4 (0.59) | 1.4 (0.86)
  20 minutes post-CAC | 1.1 (1.14) | 0.5 (0.65) | 0.4 (0.59) | 1.4 (0.87)

34. Secondary Outcome: Nasal Composite Score at Duration of Action (16 Hours Post-dose)
Description: A nasal composite score was summed for each patient based on the presence of at least one of the following four nasal symptoms on a 0-4 scale (0=none to 4=severe): rhinorrhea; nasal pruritus; ear or palate pruritus; and nasal congestion. The percentage of subjects with at least one nasal symptom present was calculated for each time point.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Number; unit: percentage of subjects
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
percentage of subjects
  7 minutes post-CAC | 82.6 | 66.7 | 52.4 | 76.0
  15 minutes post-CAC | 82.6 | 79.2 | 90.5 | 84.0
  20 minutes post-CAC | 91.3 | 83.3 | 95.2 | 84.0

35. Secondary Outcome: Nasal Composite Score at Duration of Action (24 Hours Post-dose)
Description: as for outcome 34
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Number; unit: percentage of subjects
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
percentage of subjects
  7 minutes post-CAC | 69.6 | 76.0 | 85.7 | 68.0
  15 minutes post-CAC | 82.6 | 84.0 | 90.5 | 92.0
  20 minutes post-CAC | 82.6 | 88.0 | 81.0 | 92.0

36. Secondary Outcome: Nasal Composite Score at Onset of Action (15 Minutes Post-dose)
Description: as for outcome 34
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Number; unit: percentage of subjects
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 23 | 25 | 21 | 25
percentage of subjects
  7 minutes post-CAC | 52.2 | 56 | 47.6 | 72
  15 minutes post-CAC | 82.6 | 56 | 47.6 | 84
  20 minutes post-CAC | 73.9 | 52 | 52.4 | 84

37. Secondary Outcome: Tolerability of Study Medication at Visit 3A
Description: Subjects were asked to rate the comfort of the drop in each eye upon instillation, at 1 minute, and at 2 minutes after instillation of study medication. The assessment used a 10-point scale with 0 as very comfortable and 10 as very uncomfortable. Higher scores represent a worse outcome..
Time Frame: upon instillation, 1 minute and 2 minutes post instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 25 | 26 | 25 | 25
units on a scale
  Upon instillation | 0.5 (0.95) | 0.7 (1.04) | 1.3 (1.93) | 0.6 (1.03)
  1 minute post-instillation: number analyzed (Participants) | 24 | 26 | 25 | 25
  1 minute post-instillation | 0.7 (1.13) | 0.9 (1.13) | 2.0 (2.25) | 0.9 (1.18)
  2 minutes post-instillation | 0.8 (1.10) | 1.0 (1.18) | 1.7 (2.27) | 0.6 (0.79)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion, approximately two months. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited or observed.
Arm/Group | AC-170 0.05% | AC-170 0.1% | AC-170 0.24% | AC-170 0%
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 3/26 | 4/25 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.05% (N=25) | AC-170 0.1% (N=26) | AC-170 0.24% (N=25) | AC-170 0% (N=25)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reducsed (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palatal Oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes